CLINICAL TRIAL: NCT04354883
Title: The Schmitz-Hinkelbein Method. A New Method for the Performance of External Chest Compressions During Microgravity.
Brief Title: The Schmitz-Hinkelbein Method. A New Technique for CPR in Space.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1069_1
Record Dates: First submitted 2020-04-02; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Arrest
Keywords: cardiopulmonary resuscitation; CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schmitz-Hinkelbein-Method (Active Comparator)
  Interventions: Procedure: External Chest Compressions on Manikin in Underwater Setting
- Hinkelbein-Schmitz-Method (Active Comparator)
  Interventions: Procedure: External Chest Compressions on Manikin in Underwater Setting

INTERVENTIONS:
Procedure: External Chest Compressions on Manikin in Underwater Setting — Two different methods of CPR in an analogue model of mircogravity

SUMMARY:
The risk of a severe medical event during long-duration spaceflight is significant and can endanger both the whole mission and crew. There is a certain risk for a cardiac arrest in space requiring cardiopulmonary resuscitation (CPR). So far, 5 known techniques to perform CPR in microgravity have been reported.

The aim of the present study was to describe and gather data for two new CPR techniques useful in microgravity.

DETAILED DESCRIPTION:
The risk of a severe medical event during long-duration spaceflight is significant and can endanger both the whole mission and crew. There is a certain risk for a cardiac arrest in space requiring cardiopulmonary resuscitation (CPR). So far, 5 known techniques to perform CPR in microgravity have been reported.

The aim of the present study was to describe and gather data for two new CPR techniques useful in microgravity.

The investigators conducted a randomized controlled manikin trial and asked 15 participants with valid diving-license to resuscitate a manikin in two different techniques of CPR in a free-floating position underwater. The first technique, (Schmitz-Hinkelbein-Method) is similar to conventional CPR, with the patient in a supine position on the performer's knees for stabilization. The second technique (Hinkelbein-Schmitz-Method) is similar to the first, but chest compressions are conducted with the elbow.

ELIGIBILITY:
Inclusion Criteria:

* Valid diving-license(SSI - Open Water Diver (OWD), CMAS *, PADI Open Water Diver, ISO 24801-2 (Autonomous Diver), NAUI Scuba Diver or equal license
* German EMT-qualification

Exclusion Criteria:

* any acute or chronic ENT illness/injury
* no valid diving/EMT license

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
total number of chest compressions | 60 seconds video clip with afterwards evaluation
  defined as >2 cm of compression depth
number of correct chest compressions | 60 seconds video clip with afterwards evaluation
  defined as 50-60 mm of depth
compression rate | 60 seconds video clip with afterwards evaluation
  defined as any compression of the thorax
correct compression rate | 60 seconds video clip with afterwards evaluation
  defined as 100-120 compressions min-1
depth rate | 60 seconds video clip with afterwards evaluation
  defined as 50-60 mm of depth

SECONDARY OUTCOMES:
no-flow-time | 60 seconds video clip with afterwards evaluation
  time without effective compression after the onset of chest compressions
thorax release | 60 seconds video clip with afterwards evaluation
  correct thorax release after compression
Self-Satisfaction-Score | 60 Seconds, Questionnaire filled out by participants after dive
  Depth Frequency Feasibility Exhaustion All in All Quality

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitz J, Ahlback A, DuCanto J, Kerkhoff S, Komorowski M, Low V, Russomano T, Starck C, Thierry S, Warnecke T, Hinkelbein J. Randomized Comparison of Two New Methods for Chest Compressions during CPR in Microgravity-A Manikin Study. J Clin Med. 2022 Jan 27;11(3):646. doi: 10.3390/jcm11030646. PMID 35160097